CLINICAL TRIAL: NCT03158038
Title: A Phase 4 Randomized, Double-blind, Placebo-controlled Study to Evaluate the Safety of 1 New 6:2 Influenza Virus Reassortant in Adults
Brief Title: Study to Evaluate the Safety of 1 New 6:2 Influenza Virus Reassortant in Adults for the 2017-2018 Season
Acronym: FluMist
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: MedImmune LLC (Industry)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: D2560C00014
Record Dates: First submitted 2017-05-16; First posted 2017-05-17 (Actual); Results first posted 2019-01-04 (Actual); Last update posted 2019-01-04 (Actual); Status verified 2018-12

CONDITIONS: Influenza; Healthy
Keywords: Trivalent; Influenza; FluMist Quadrivalent; Vaccine; Prevention; Healthy; Monovalent
MeSH Terms: conditions — Influenza, Human | interventions — Influenza Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Monovalent Influenza Vaccine (Experimental): Participants will receive a single dose of monovalent influenza vaccine [10^7.0 +/- 0.5 fluorescent focus unit (FFU) of each of 1 cold adapted (ca), attenuated (att), temperature sensitive (ts) 6:2 reassortant influenza strain] by intranasal spray on Day 1.
  Interventions: Biological: Monovalent Influenza Vaccine
- Placebo (Placebo Comparator): Participants will receive a single dose of placebo matching with monovalent influenza vaccine by intranasal spray on Day 1.
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Monovalent Influenza Vaccine — A single dose of monovalent influenza vaccine [10^7.0 +/- 0.5 FFU of each of 1 ca, att, ts 6:2 reassortant influenza strain] will be administered as intranasal spray on Day 1.
  Arms: Monovalent Influenza Vaccine
Other: Placebo — A single dose of placebo matching with monovalent influenza vaccine will be administered as intranasal spray on Day 1.
  Arms: Placebo

SUMMARY:
This prospective annual release study is designed to evaluate the safety of 1 new influenza virus vaccine strain to be included in FluMist Quadrivalent for the 2017-2018 influenza season.

DETAILED DESCRIPTION:
This prospective, randomized, double-blind, placebo-controlled release study will enroll approximately 300 healthy adults 18 to 49 years of age (not yet reached their 50th birthday). Eligible participants will be randomly assigned in a 4:1 fashion to receive a single dose of monovalent vaccine or placebo by intranasal spray. Randomization will be stratified by site. This study will be conducted at 2 sites in the United States of America. Each participant will receive 1 dose of investigational product on Day 1. The duration of study participation for each participant is the time from study vaccination through 180 days after study vaccination.

ELIGIBILITY:
Key Inclusion Criteria:

* Age 18 through 49 years
* Written informed consent
* Participant available by telephone
* Ability to understand and comply with the requirements of the protocol, as judged by the Investigator

Key Exclusion Criteria:

* Concurrent enrollment in another clinical study up to 180 days after receipt of investigational product (Day 181)
* History of hypersensitivity to any component of the vaccine, including egg or egg protein or serious, life threatening, or severe reactions to previous influenza vaccinations
* Any condition for which the inactivated influenza vaccine is indicated, including chronic disorders of the pulmonary or cardiovascular systems (example [eg], asthma), chronic metabolic diseases (eg, diabetes mellitus), renal dysfunction, or hemoglobinopathies that required regular medical follow-up or hospitalization during the preceding year
* Acute febrile (greater than [>] 100.0 degrees Fahrenheit [F] oral or equivalent) and/or clinically significant respiratory illness (example, cough or sore throat) within 14 days to randomization
* Any known immunosuppressive condition or immune deficiency diseases, including human immunodeficiency virus infection, or ongoing immunosuppressive therapy
* History of Guillain-Barre syndrome
* Receipt of any investigational agent within 30 days prior to randomization, or expected receipt through 30 days after the dose of investigational product (use of licensed agents for indications not listed in the Package Insert is permitted)
* Receipt of any non-study vaccine within 30 days prior to randomization, or expected receipt through 30 days after receipt of investigational product
* Expected receipt of antipyretic or analgesic medication on a daily or every other day basis from randomization through 14 days after receipt of investigational product
* Administration of intranasal medications within 14 days prior to randomization, or expected receipt through 14 days after administration of investigational product
* Receipt of influenza antiviral therapy or influenza antiviral agents within 48 hours prior to investigational product administration or expected receipt of influenza antiviral therapy or influenza antiviral agents through 14 days after receipt of investigational product

Ages: 18 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 300 (Actual)
Dates: Start 2017-05-30 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Research Site, Stockbridge, Georgia
  - Research Site, Portland, Oregon

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted from 30 May 2017 to 14 Dec 2017 at 2 sites in the United States of America (USA).
Pre-assignment Details: A total of 300 participants were randomized and participated in the study.
Groups:
- Monovalent Influenza Vaccine: Participants received a single dose of monovalent influenza vaccine [10^7.0 +/- 0.5 fluorescent focus unit (FFU) of each of 1 cold adapted (ca), attenuated (att), temperature sensitive (ts) 6:2 reassortant influenza strain] by intranasal spray on Day 1.
- Placebo: Participants received a single dose of placebo matching with monovalent influenza vaccine by intranasal spray on Day 1.
Period: Overall Study
Arm/Group | Monovalent Influenza Vaccine | Placebo
Started | 240 | 60
Completed | 240 | 60
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: The intent-to-treat (ITT) population included all participants who were randomized and treated with investigational product.
Groups:
- Total: Total of all reporting groups
Arm/Group | Monovalent Influenza Vaccine | Placebo | Total
Number analyzed (Participants) | 240 | 60 | 300
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: The ITT population included all participants who were randomized and treated with investigational product.
  Years | 29.9 (9.5) | 32.5 (10.5) | 30.4 (9.8)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: The ITT population included all participants who were randomized and treated with investigational product.
  Participants
    Female | 138 | 33 | 171
    Male | 102 | 27 | 129
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ITT population included all participants who were randomized and treated with investigational product.
  Participants
    Hispanic or Latino | 13 | 3 | 16
    Not Hispanic or Latino | 227 | 57 | 284
    Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: The ITT population included all participants who were randomized and treated with investigational product.
  Participants
    American Indian or Alaska Native | 1 | 0 | 1
    Asian | 3 | 1 | 4
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
    Black or African American | 36 | 6 | 42
    White | 191 | 52 | 243
    More than one race | 8 | 1 | 9
    Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Fever Greater Than or Equal to (>=) 101 Degrees Fahrenheit (F)
Description: Percentage of participants with fever defined as oral temperature >=101 degrees F were reported.
Time Frame: Baseline (Day 1) up to Day 8
Population: as for baseline characteristics
Measure: Number; unit: Percentage of Participants
Groups:
- Monovalent Influenza Vaccine: Participants received a single dose of monovalent influenza vaccine [10^7.0 +/- 0.5 fluorescent focus unit (FFU) of each of 1 cold adapted (ca), attenuated (att), temperature sensitive (ts) 6:2 reassortant influenza strains] by intranasal spray on Day 1.
Arm/Group | Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Percentage of Participants | 0 | 0
Statistical Analysis 1: Comparison: Monovalent Influenza Vaccine vs Placebo; Test type: Superiority; Rate difference = 0, 95% CI 2-sided [-6.7 to 1.9]

2. Secondary Outcome: Percentage of Participants With Solicited Symptoms
Description: Solicited symptoms are predefined symptoms or events specifically inquired about and assessed daily after vaccine administration up to 15 days after vaccination. The solicited symptoms include fever greater than (>) 100.0 degrees F (37.8 degrees Celsius), runny nose, sore throat, cough, vomiting, muscle aches, chills, decreased activity and headache. Results were reported for all solicited symptoms except fever >=101 degrees F (reported as primary outcome) up to 8 days after vaccination and all solicited symptoms up to 15 days after vaccination.
Time Frame: Baseline (Day 1) up to Day 8 and Day 15
Population: The ITT population included all participants who were randomized and treated with investigational product.
Measure: Number; unit: Percentage of Participants
Arm/Group | Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Percentage of Participants
  Up to Day 8 | 27.9 | 26.7
  Up to Day 15 | 32.1 | 31.7
Statistical Analysis 1: Comparison: Monovalent Influenza Vaccine vs Placebo; Statistical analysis up to Day 8; Test type: Superiority; Rate difference = 1.3, 95% CI 2-sided [-12.8 to 13.2]
Statistical Analysis 2: Comparison: Monovalent Influenza Vaccine vs Placebo; Statistical analysis up to Day 15; Test type: Superiority; Rate difference = 0.4, 95% CI 2-sided [-14.1 to 13.2]

3. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent AEs were events between administration of study drug and up to 15 days after vaccination that are absent before treatment or that worsened relative to pre-treatment state. Results were given for AEs reported up to 8 days and 15 days after vaccination.
Time Frame: Baseline (Day 1) up to Day 8 and Day 15
Population: The ITT population included all participants who were randomized and treated with investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Participants
  Up to Day 8 | 13 | 0
  Up to Day 15 | 19 | 1

4. Secondary Outcome: Number of Participants With Treatment-Emergent Serious Adverse Events (TESAEs) and New Onset Chronic Diseases (NOCDs)
Description: An AE is any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An serious adverse event (SAE) is an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent SAEs were serious events between administration of study drug and up to 181 days after the dose that are absent before treatment or that worsen relative to pretreatment state. An NOCD is a newly diagnosed medical condition that is of a chronic, ongoing nature and is assessed by the investigator as medically significant. Results were given for TESAEs and NOCDs reported up to 29 days and 181 days after vaccination.
Time Frame: Baseline (Day 1) up to Day 29 and Day 181
Population: The ITT population included all participants who were randomized and treated with investigational product.
Measure: Count of Participants; unit: Participants
Arm/Group | Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Participants
  TESAEs: Up to Day 29 | 1 | 0
  NOCDs: Up to Day 29 | 0 | 0
  TESAEs: Up to Day 181 | 1 | 0
  NOCDs: Up to Day 181 | 1 | 0

5. Secondary Outcome: Percentage of Participants Who Require Antipyretic and/or Analgesic Medication
Description: Percentage of participants who require antipyretic and/or analgesic medication were reported.
Time Frame: Baseline (Day 1) up to Day 8 and Day 15
Population: The ITT population included all participants who were randomized and treated with investigational product.
Measure: Number; unit: Percentage of participants
Arm/Group | Monovalent Influenza Vaccine | Placebo
Number analyzed (Participants) | 240 | 60
Percentage of participants
  Up to Day 8 | 2.1 | 1.7
  Up to Day 15 | 3.3 | 6.7

ADVERSE EVENTS:
Time Frame: Adverse Events: Baseline (Day 1) up to Day 15, and Serious Adverse Events: Baseline (Day 1) up to Day 181
Arm/Group | Monovalent Influenza Vaccine | Placebo
All-Cause Mortality (participants affected / at risk) | 0/240 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/240 | 0/60
Other Adverse Events (participants affected / at risk) | 19/240 | 1/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monovalent Influenza Vaccine (N=240) | Placebo (N=60)
Endometriosis (Reproductive system and breast disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Monovalent Influenza Vaccine (N=240) | Placebo (N=60)
Ear congestion (Ear and labyrinth disorders) | 1 | 0
Ear pain (Ear and labyrinth disorders) | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Ear infection (Infections and infestations) | 1 | 0
Laryngitis (Infections and infestations) | 2 | 0
Viral infection (Infections and infestations) | 0 | 1
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 1 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 0
Nasal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Sneezing (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
MedImmune has 60 days to review results communications prior to public release and may delete information that compromises on-going studies or is considered proprietary. This restriction is not intended to compromise the objective scientific integrity of the manuscript, it being understood that results shall be published regardless of outcome.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-03-03): https://cdn.clinicaltrials.gov/large-docs/38/NCT03158038/Prot_SAP_000.pdf